CLINICAL TRIAL: NCT05214872
Title: Assessment of the Impact of Selected Factors on the Cardiovascular System in Patients With Different Chronic Kidney Disease Stages
Brief Title: The Impact of Selected Factors on the Cardiovascular System in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dorota Formanowicz, MD.Ph.D. Associate Professor, Poznan University of Medical Sciences
Other Study IDs: PoznanUMS_DF2
Record Dates: First submitted 2021-12-09; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Atherosclerosis of Artery; Inflammation; Chronic Kidney Diseases; Dialysis; Complications; Cardiovascular Diseases
Keywords: risk factors; chronic kidney disease; inflammation; oxidative stress; atherosclerosis; mortality
MeSH Terms: conditions — Inflammation; Renal Insufficiency, Chronic; Cardiovascular Diseases; Atherosclerosis | interventions — Body Mass Index; Carotid Intima-Media Thickness; Blood Circulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- PREDIALYSIS GROUP: (n = 48) - patients in the pre-dialysis period (stages G3b-G4 of chronic kidey disease (CKD)) with moderate or severe decrease in estimated glomerular filtration rate (eGFR) (eGFR 44-29 ml/min/1.73 m^2)
  Interventions: Diagnostic Test: laboratory parameters - complete blood count; Other: body mass index (BMI) [kg/m^2] calculation; Diagnostic Test: selected parameters of oxidative stress (1); Diagnostic Test: metalloproteinases; Diagnostic Test: parameters of lipids metabolism in the serum; Diagnostic Test: parameters of iron metabolism; Diagnostic Test: selected inflammatory markers; Device: carotid intima-media thickness (IMT); Device: non-invasive cardiological examinations; Device: vessel stiffness assessment; Other: cardiovascular (CV)-related death recording during 2-year follow-up; Diagnostic Test: glucose (Glu); Diagnostic Test: klotho; Diagnostic Test: fibroblast growth factor 23 (FGF-23); Diagnostic Test: parameters of calcium and phosphate metabolism; Diagnostic Test: liver enzymes activity assessment; Diagnostic Test: total protein and albumin; Diagnostic Test: creatinine and urea; Diagnostic Test: selected parameters of oxidative stress (2); Diagnostic Test: selected parameters of oxidative stress (3) sRAGE; Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups; Diagnostic Test: selected electrolytes assessment; Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP); Other: estimated glomerular filtration rate (eGFR) calculation
- END-STAGE RENAL DISEASE (ESRD) GROUP: Patients with ESRD (n=106) - (eGFR <15 ml/min /1.73 m^2) undergoing renal replacement therapy have formed this group.
  Depending on the method of renal replacement therapy used, two subgroups have been distinguished: (1) peritoneal dialysis (PD) subgroup (n=35) including patients treated by peritoneal dialysis. In this subgroup, due to the treatment technique, two groups have been distinguished, a group (n=15) treated with the automatic peritoneal dialysis (APD) technique and a group (n = 20) using the technique of continuous cycling peritoneal dialysis (CCPD), (2) hemodialysis (HD) subgroup (n = 71) including patients treated with repeated hemodialysis. The duration of hemodialysis was at least 10 hours/week using standard bicarbonate dialysis fluids and polysulfone low-flux dialyzers. The blood flow during hemodialysis was 200-350 ml/min, with an average dialysis fluid flow of 500 ml/min.
  Interventions: Diagnostic Test: laboratory parameters - complete blood count; Other: body mass index (BMI) [kg/m^2] calculation; Diagnostic Test: selected parameters of oxidative stress (1); Diagnostic Test: metalloproteinases; Diagnostic Test: parameters of lipids metabolism in the serum; Diagnostic Test: parameters of iron metabolism; Diagnostic Test: selected inflammatory markers; Device: carotid intima-media thickness (IMT); Device: non-invasive cardiological examinations; Device: vessel stiffness assessment; Other: cardiovascular (CV)-related death recording during 2-year follow-up; Diagnostic Test: glucose (Glu); Diagnostic Test: klotho; Diagnostic Test: fibroblast growth factor 23 (FGF-23); Diagnostic Test: parameters of calcium and phosphate metabolism; Diagnostic Test: liver enzymes activity assessment; Diagnostic Test: total protein and albumin; Diagnostic Test: creatinine and urea; Diagnostic Test: selected parameters of oxidative stress (2); Diagnostic Test: selected parameters of oxidative stress (3) sRAGE; Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups; Diagnostic Test: selected electrolytes assessment; Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP); Other: estimated glomerular filtration rate (eGFR) calculation
- CARDIOLOGY (CARD) GROUP: CARD group (n = 37) - patients with at least one history of a cardiovascular event, admitted to hospital for elective angiography, without any signs of impaired kidney function.
  The studies in this group were conducted to check the changes that occur as a result of cardiovascular disease (CVD) but without kidney disease.
  Interventions: Diagnostic Test: laboratory parameters - complete blood count; Other: body mass index (BMI) [kg/m^2] calculation; Diagnostic Test: selected parameters of oxidative stress (1); Diagnostic Test: metalloproteinases; Diagnostic Test: parameters of lipids metabolism in the serum; Diagnostic Test: parameters of iron metabolism; Diagnostic Test: selected inflammatory markers; Device: carotid intima-media thickness (IMT); Device: non-invasive cardiological examinations; Device: vessel stiffness assessment; Other: cardiovascular (CV)-related death recording during 2-year follow-up; Diagnostic Test: glucose (Glu); Diagnostic Test: klotho; Diagnostic Test: fibroblast growth factor 23 (FGF-23); Diagnostic Test: parameters of calcium and phosphate metabolism; Diagnostic Test: liver enzymes activity assessment; Diagnostic Test: total protein and albumin; Diagnostic Test: creatinine and urea; Diagnostic Test: selected parameters of oxidative stress (2); Diagnostic Test: selected parameters of oxidative stress (3) sRAGE; Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups; Diagnostic Test: selected electrolytes assessment; Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP); Other: estimated glomerular filtration rate (eGFR) calculation
- Chronic kidney disease (CKD) 1-2 GROUP: CKD1-2 (n=29) (stage G1-G2 CKD) with mild decrease in eGFR (eGFR >90-60 ml/min/1.73 m^2)
  The studies in this group were performed to disclose the changes that occur as a consequence of the beginning of kidney function deterioration.
  Interventions: Diagnostic Test: laboratory parameters - complete blood count; Other: body mass index (BMI) [kg/m^2] calculation; Diagnostic Test: selected parameters of oxidative stress (1); Diagnostic Test: metalloproteinases; Diagnostic Test: parameters of lipids metabolism in the serum; Diagnostic Test: parameters of iron metabolism; Diagnostic Test: selected inflammatory markers; Device: carotid intima-media thickness (IMT); Device: non-invasive cardiological examinations; Device: vessel stiffness assessment; Other: cardiovascular (CV)-related death recording during 2-year follow-up; Diagnostic Test: glucose (Glu); Diagnostic Test: klotho; Diagnostic Test: fibroblast growth factor 23 (FGF-23); Diagnostic Test: parameters of calcium and phosphate metabolism; Diagnostic Test: liver enzymes activity assessment; Diagnostic Test: total protein and albumin; Diagnostic Test: creatinine and urea; Diagnostic Test: selected parameters of oxidative stress (2); Diagnostic Test: selected parameters of oxidative stress (3) sRAGE; Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups; Diagnostic Test: selected electrolytes assessment; Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP); Other: estimated glomerular filtration rate (eGFR) calculation
- Healthy volunteers (HV): HV (n = 32) - this group was composed of healthy people, with no evidence of impairment in renal function and cardiovascular disorders in the history and at the time of enrollment in the study.
  Interventions: Diagnostic Test: laboratory parameters - complete blood count; Other: body mass index (BMI) [kg/m^2] calculation; Diagnostic Test: selected parameters of oxidative stress (1); Diagnostic Test: metalloproteinases; Diagnostic Test: parameters of lipids metabolism in the serum; Diagnostic Test: parameters of iron metabolism; Diagnostic Test: selected inflammatory markers; Device: carotid intima-media thickness (IMT); Device: non-invasive cardiological examinations; Device: vessel stiffness assessment; Other: cardiovascular (CV)-related death recording during 2-year follow-up; Diagnostic Test: glucose (Glu); Diagnostic Test: klotho; Diagnostic Test: fibroblast growth factor 23 (FGF-23); Diagnostic Test: parameters of calcium and phosphate metabolism; Diagnostic Test: liver enzymes activity assessment; Diagnostic Test: total protein and albumin; Diagnostic Test: creatinine and urea; Diagnostic Test: selected parameters of oxidative stress (2); Diagnostic Test: selected parameters of oxidative stress (3) sRAGE; Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups; Diagnostic Test: selected electrolytes assessment; Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP); Other: estimated glomerular filtration rate (eGFR) calculation

INTERVENTIONS:
Diagnostic Test: laboratory parameters - complete blood count — the complete blood count was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA):
  * hemoglobin (HGB) [g/dl];
  * red blood count (RBC) [10^12/l];
  * hematocrit (HCT) [l/l];
  * white blood cells (WBC) [10^9/l];
  * platelet count (PLT) [10^9/l]
Other: body mass index (BMI) [kg/m^2] calculation — body mass index (BMI) [kg/m^2] was calculated by dividing a person's weight (post-HD weight in HD group) [kg] by the squared their body height [m]
Diagnostic Test: selected parameters of oxidative stress (1) — Serum concentration of:
  * advanced glycation ends products (AGE) [µg/mg protein];
  * 3-nitrotyrosine (3-NT) [µmol/mg protein];
  * advanced oxidation protein products (AOPP) [µmol/mg protein];
  * carboxymethyle(lysine) (CML) [µg/mg protein]
  were determined with the enzyme immunoassay methods (ELISA) using Shanghai Sunred Biological Technology Co kits, China.
Diagnostic Test: metalloproteinases — metalloproteinases in the serum [ng/ml]:
  * metalloproteinase 9 (MMP-9) in the serum was determined by the ELISA method using the Quantikine Human MMP-9 (total) kit, by R&D Systems, Canada;
  * tissue inhibitor of metalloproteinase 1 (TIMP-1) in the serum - was determined by the ELISA method using the Quantikine Human TIMP-1 kit, manufactured by R&D Systems, Canada;
  * the MMP-9/TIMP-1 ratio was calculated by the quotient of the MMP-9 and the TIMP-1 concentration.
Diagnostic Test: parameters of lipids metabolism in the serum — * total cholesterol (T-C) [mg/dl] - was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA;
  * low-density lipoprotein cholesterol (LDL-C) [mg/dl] - was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA;
  * high-density lipoprotein cholesterol (HDL-C) [mg/dl] - was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA;
  * triglycerides (TG) [mg/dl] - were assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA;
  * the concentration of low-density lipoprotein (LDL-C) cholesterol - was determined from Friedewalds' equation (LDL-C [mg/dl] = total cholesterol (T-C) [mg/dl]- HDL-C [mg/dl]- TG[mg/dl]/5).
Diagnostic Test: parameters of iron metabolism — * iron concentration [mg/dl] - was analyzed with the Cobas Integra 400 plus biochemical analyzer from Roche Diagnostics, USA;
  * total iron-binding capacity (TIBC) [mg/dl] - was analyzed with the Cobas Integra 400 plus biochemical analyzer from Roche Diagnostics, USA;
  * the unsaturated iron-binding capacity (UIBC) [mg/dl] was determined by an equation in which iron concentration in plasma is subtracted from TIBC [mg/dl];
  * ferritin [ng/ml] concentration was determined with the Modular E-170 biochemical analyzer from Roche Diagnostics, USA.
Diagnostic Test: selected inflammatory markers — * high-sensitivity C-reactive protein (hsCRP) [mg/l] was measured using DADE Behring, USA and the DADE nephelometer Behring Analyzer II;
  * neopterin [nmol/l] was determined by using the Neopterin ELISA kit, DRG International, Inc., USA;
  * interleukin 18 (IL-18) [pg/ml] concentration was determined by Colorimetric Sandwich ELISA, Quantikine Human IL-18 R&D Inc., USA.
Device: carotid intima-media thickness (IMT) — carotid intima-media thickness (IMT) [mm] was measured by The Accuson CV 70 system (Siemens) with a 10 megahertz (Mhz) transducer.
  Two longitudinal projections were assessed (anterolateral and posterolateral). The distal 1 cm of the common carotid artery just proximal to the bulb was measured by means of a computer analysis system (Medical Imaging Applications, LLC).
Device: non-invasive cardiological examinations — For non-invasive cardiological examinations, the Portapres device (Finapres Medical Systems (FMS), the Netherlands), the SphygmoCor tonometer (AtCor Medical), the Colin blood pressure monitor (BMP)-7000 (Japan) were used.
  Main assessed variables: heart rate (HR) [beats per minute [bpm]]; ejection duration (ED) [millisecons]; peripheral systolic (pSBP) and diastolic blood pressure (pDBP) [mm Hg]; peripheral mean arterial pressure (pMAP) [mm Hg]; peripheral end-systolic pressure (pESP) [mm Hg]; central systolic (cSBP) and diastolic blood pressure (cDBP) [mm Hg]; central mean arterial pressure (cMAP) [mm Hg]; central augmented pressure (cAP) [mmHg]; central mean pressure of diastole (cMPD)[mm Hg]; central mean pressure of systole (cMPS) [mm Hg]; central end-systolic pressure (cESP) [mm Hg].
Device: vessel stiffness assessment — The following parameters of vessel stiffness were assessed by Pulse Trace 2000 (Micro Medical Ltd., Rochester, Kent, United Kingdom):
  * reflection index (RI) [in percentages [%]];
  * vascular stiffness index (SI) [m/s];
  * peripheral pulse pressure (pPP) [mm Hg];
  * central puls pressure (cPP) [mm Hg]
  * peripheral pulse pressure/central pulse pressure (pPP/cPP ratio).
Other: cardiovascular (CV)-related death recording during 2-year follow-up — During a 2-year follow-up from the enrollment to this study, CV-related fatal incidents history has been recorded for each subject separately. The primary endpoint was fatal acute myocardial infarction (AMI) or acute ischemic stroke or any unexpected or sudden death only if autopsy proved CV-related. If there was doubt about the cause of death or there was no contact with the patient during the two years from study enrollment, that patient was excluded and not considered further.
Diagnostic Test: glucose (Glu) — glucose (Glu) [mg/dl] was assessed in the serum by a routine technique using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: klotho — klotho [ng/ml] - was analyzed in the serum by Human KL(Klotho) [ng/ml] ELISA Kit, Shanghai Sunred Biological Technology Co kit, China.
Diagnostic Test: fibroblast growth factor 23 (FGF-23) — FGF-23 [pg/ml] - was analyzed in rhe serum using Human FGF-23 ELISA Kit, Sigma-Aldrich, USA.
Diagnostic Test: parameters of calcium and phosphate metabolism — * total and ionized calcium [mg/dl],
  * phosphate [mg/dl],
  * intact parathormone (iPTH) [mg/dl]
  were assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: liver enzymes activity assessment — activity of:
  * alanine transaminase (ALT) [U/l];
  * aspartate transaminase (AST) [U/l];
  * alkaline phosphatase (ALP) [U/l]
  were assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: total protein and albumin — * total protein (TP) [g/dl];
  * albumin (ALB) [g/dl]
  were assessed in the serum by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: creatinine and urea — * creatinine in the serum [mg/dl] - the assay is based on the reaction of creatinine with sodium picrate as described by Jaffe (Jaffes' colorimetric method) - was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA;
  * urea [mg/dl] in the serum - was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: selected parameters of oxidative stress (2) — myeloperoxidase (MPO) [ng/ml] in the serum- was determined by the ELISA method using the Quantikine Human MPO test by R&D Systems kit, Canada.
Diagnostic Test: selected parameters of oxidative stress (3) sRAGE — soluble receptor for advanced glycation end products (sRAGE) [µg/mg protein] in the serum was tested with enzymatic immunoassay (Quantikine ELISA) using R&D Systems kit, Canada.
Diagnostic Test: selected parameters of oxidative stress (4) MG, CEL, carbamyl protein groups — * methylglyoxal (MG) [µg/mg protein];
  * carboxyethyle(lysine) (CEL) [µg/mg protein];
  * carbamyl protein groups [µg/mg protein] were assessed in the serum by competitive enzyme immunoassay (competitive ELISA) using kits from Cell Biolabs Inc, USA.
Diagnostic Test: selected electrolytes assessment — * potassium (K) [mmol/l];
  * sodium (Na) [mmol/l];
  * magnesium (Mg) [mg/dL]
  were assessed in the serum by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic Test: NT-pro-brain natriuretic peptide (NT-proBNP) — NT-proBNP [fmol/ml] - was analyzed in the serum by enzyme immunoassay using the Nt-proBNP kit from Biomedica, Slovakia.
Other: estimated glomerular filtration rate (eGFR) calculation — eGFR [ml/min/1.73m^2] - according to the Kidney Disease: Improving Global Outcomes (KDIGO) 2012 recommendations was calculated based on the Modification of Diet in Renal Disease (MDRD) formula: eGFR = 186 x [creatinine concentration in mg/dl] - 1.154 x [age in years] - 0.203 x [0.724] for the female gender.

SUMMARY:
Chronic kidney disease (CKD), is characterized by accelerated development of atherosclerosis and advanced remodelling of vessels and the heart. It is associated with many factors, including inflammation, arterial hypertension, hyperlipidemia, hyperhomocysteinemia, secondary hyperparathyroidism, and oxidative stress. Hypertension is one of the most critical risk factors for cardiovascular complications. It leads to the formation of structural changes in the vascular system: it impairs the activity of the endothelium, causes hypertrophy and remodelling of the vascular wall, reduces the susceptibility of the vessels and accelerates the development of atherosclerosis. This study aimed to identify the processes and their representative markers, the concentration of which in the serum may reflect the cardiovascular system status and can predict the increased mortality in HD patients.

DETAILED DESCRIPTION:
Chronic Kidney Disease has a significant impact on the cardiovascular system. From many different complications of CKD, one to mention is arterial stiffness. This disorder results from many pathologies, including inflammation, arterial hypertension, carbohydrate metabolic disorders, lipid disorders, vascular calcification, chronic inflammation, and oxidative stress.

The main goal of this study was to analyze the mechanisms leading to the increased tendency to cardiovascular disturbances in CKD, with particular focus on the parameters of oxidative stress, inflammation and the results of imaging examinations (intima-media thickness (IMT) assessments) and other non-invasive cardiological examinations based on the results using the Portapres device (Finapres Medical Systems (FMS), the Netherlands), the SphygmoCor tonometer (AtCor Medical), the Colin blood pressure monitor (BMP)-7000 (Japan) Pulse Trace 2000 (Micro Medical Ltd., Rochester, Kent, United Kingdom) The Accuson CV 70 system (Siemens) with a 10 megahertz (Mhz) transducer.

Besides, studied participants were followed 2 years after enrollment to study for recording cardiovascular-related death.

ELIGIBILITY:
Criteria:

The following criteria of qualifying for the study were adopted for all respondents:

* 18 years of age or older,
* written consent to participate in the study,
* no active inflammatory process,
* no neoplastic disease or a neoplastic disease whose treatment was stopped at least 10 years ago,
* no history of immunosuppressive treatment,
* stable liver function (not more than two times increased activity of transaminases), HBs antigen and anti-HCV negative antibodies,anti-HIV negative antibodies.

In addition, for CKD patients (CKD1-2) and PREDIALYSIS GROUP, the following additional inclusion conditions were applied:

* no acute cardiovascular complications, ie acute heart failure, hypertensive crisis, acute coronary syndrome, at the time of study entry.

At the same time, depending on the technique of renal replacement therapy used, additional inclusion criteria were established for each of the subgroups:

in group HD:

* a minimum of 6 months of treatment with repeated hemodialysis, 3 times a week, for a minimum of 10 hours a week,
* arteriovenous fistula as a vascular access for hemodialysis,
* Estimated dialysis adequacy ratio (eKt / V) of at least 1.2. in the PD group:
* treatment duration UP to a minimum of 6 months, Kt / V ≥1.8 l / week / 1.73 m2.

For CARD patients, additional conditions include:

* no obvious evidence of renal impairment in the history and at the time of study entry, renal function assessed on the basis of eGFR and urine albumin/creatinine ratio,
* history of angina pectoris,
* documented history of at least one acute coronary syndrome,
* admission to the Department of Intensive Care of Cardiology and Internal Diseases in order to perform a planned coronary angiography, on the day of admission to the study without signs of the acute coronary syndrome, no additional comorbidities, ie those that do not result directly or indirectly from coronary heart disease.

In turn, for the HV group (control group), additional conditions include:

* no obvious evidence of renal impairment in the history and at the time of study entry, renal function assessed on the basis of eGFR and urine albumin/creatinine ratio,
* no obvious signs of cardiovascular impairment in the history and at the time of study entry, estimated on the basis of normal blood pressure (<140/90 mmHg), no abnormalities in the medical history and physical examination,
* not taking any medications on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 252 people have been enrolled on the study, including 106 consecutive dialyzed patients (HD group), treated in 2016-2018 at the Nephrology Outpatient Clinic and the Clinical Hospital's Dialysis Center. H. Święcickiego in Poznań; 37 32 healthy participants (control group), serving as a comparative group.
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic test: basic biochemical parameters: complete blood count - hemoglobin (HGB) | 3 years
  hemoglobin (HGB) [g/dl] was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA).
Diagnostic test: basic biochemical parameters: complete blood count - red blood cell count (RBC) | 3 years
  red blood cell count (RBC) [10^12/l] was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA).
Diagnostic test: basic biochemical parameters: complete blood count - hematocrit (HCT) | 3 years
  hematocrit (HCT) [l/l] was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA).
Diagnostic test: basic biochemical parameters: complete blood count - white blood cell count (WBC) | 3 years
  white blood cells (WBC) [10^9/l] was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA).
Diagnostic test: basic biochemical parameters: complete blood count - platelet count (PLT) | 3 years
  platelet count (PLT) [10^9/l] was analyzed using Sysmex K-4500 Automated Hematology Analyzer (by GMI Inc., USA).
Diagnostic test: glucose (Glu) | 3 years
  glucose (Glu) [mg/dl] concentration in the serum was assessed by the routine technique using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: urea | 3 years
  urea [mg/dl] concentration in the serum was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: creatinine | 3 years
  creatinine [mg/dl] concentration in the serum was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA (based on Jaffes' colorimetric method - the assay is based on the reaction of creatinine with sodium picrate as described by Jaffe).
Estimated glomerular filtration rate (eGFR) [ml/min/1.73m^2] calculation | 3 years
  eGFR - according to the Kidney Disease: Improving Global Outcomes (KDIGO) 2012 recommendations was calculated based on the Modification of Diet in Renal Disease (MDRD) formula: eGFR = 186 x [creatinine concentration in mg/dl] - 1.154 x [age in years] - 0.203 x [0.724] for the female gender.
Body mass index (BMI) [kg/m^2] calculation | 3 years
  Body mass index (BMI) - [kg/m^2] was calculated by dividing a person's weight (post-HD weight in HD group) [kg] by the squared their body height [m].
Diagnostic test: parameters of lipids metabolism in the serum - total cholesterol (T-C) | 3 years
  total cholesterol (T-C) [mg/dl] concentration in the serum was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: parameters of lipids metabolism in the serum - high-density lipoprotein cholesterol (HDL-C) | 3 years
  high-density lipoprotein cholesterol (HDL-C) [mg/dl] concentration in the serum was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: parameters of lipids metabolism in the serum low-density lipoprotein cholesterol (LDL-C). | 3 years
  low-density lipoprotein (LDL-C) cholesterol concentration in the serum was determined from Friedewals' equation (LDL-C [mg/dl] = total cholesterol (T-C) [mg/dl] - HDL-C [mg/dl] - TG[mg/dl]/5).
  It was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: parameters of lipids metabolism in the serum - triglycerides (TG) | 3 years
  triglycerides (TG) [mg/dl] concentration in the serum was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: liver enzymes activity assessment - aspartate transaminase (AST) | 3 years
  activity of aspartate transaminase (AST) [U/l]; was assessed in the serum by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: liver enzymes activity assessment - alanine transaminase (ALT) | 3 years
  activity of alanine transaminase (ALT) [U/l] was assessed in the serum by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: liver enzymes activity assessment - alkaline phosphatase (ALP) [U/l] | 3 years
  activity of alkaline phosphatase (ALP) [U/l] was assessed in the serum by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: total protein (TP) | 3 years
  total protein (TP) [g/dl] concentration in the serum was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: albumin(ALB) | 3 years
  albumin (ALB) [g/dl] concentration in the serum was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: parameters of iron metabolism - iron | 3 years
  iron concentration [mg/dl] in the serum - was assessed with the Cobas Integra 400 plus biochemical analyzer from Roche Diagnostics, USA;
Diagnostic test: parameters of iron metabolism - total iron-binding capacity (TIBC) | 3 years
  total iron-binding capacity (TIBC) [mg/dl] - was determined with the Cobas Integra 400 plus biochemical analyzer from Roche Diagnostics, USA.
Diagnostic test: parameters of iron metabolism - the unsaturated iron-binding capacity (UIBC) | 3 years
  unsaturated iron-binding capacity (UIBC) [mg/dl] was determined by an equation in which iron [mg/dl] concentration in plasma is subtracted from TIBC [mg/dl].
Diagnostic test: parameters of iron metabolism - ferritin | 3 years
  ferritin [ng/ml] concentration in the serum was determined with the Modular E-170 biochemical analyzer from Roche Diagnostics, USA.
Diagnostic test: total and ionized calcium | 3 years
  total and ionized calcium [mg/dl] serum concentrations were assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: phosphate | 3 years
  phosphate [mg/dl] serum concentration was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: intact parathormone (iPTH) | 3 years
  intact parathormone (iPTH) [mg/dl] serum concentration was assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: klotho (KL) | 3 years
  klotho (KL) [ng/ml] serum concentration was analyzed by Human KL(Klotho) [ng/ml] ELISA Kit, Shanghai Sunred Biological Technology Co kit, China.
Diagnostic test: fibroblast growth factor 23 (FGF-23) | 3 years
  fibroblast growth factor 23 (FGF-23) [pg/ml] serum concentration was analyzed using Human FGF-23 ELISA Kit, Sigma-Aldrich, USA.
Diagnostic test: selected electrolytes assessment in the serum: potassium (K) and sodium (Na) | 3 years
  Electrolytes: potassium (K) [mmol/l] and sodium (Na) [mmol/l] serum concentrations were assessed by the routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: selected electrolytes assessment in the serum: magnesium | 3 years
  magnesium (Mg) [mg/dl] serum concentration was assessed by routine techniques using Cobas Integra 400 plus biochemical analyzer by Roche Diagnostics, USA.
Diagnostic test: selected parameters of oxidative stress - 3-nitrotyrosine (3-NT) | 3 years
  Serum concentration of 3-nitrotyrosine (3-NT) [µmol/mg protein] was determined with the enzyme immunoassay method (ELISA) for 3NT using Shanghai Sunred Biological Technology Co kits, China.
Diagnostic test: selected parameters of oxidative stress - advanced glycation ends products (AGE) | 3 years
  Serum concentration of advanced glycation ends products (AGE) [µg/mg protein] was determined with the enzyme immunoassay method (ELISA) for AGE using Shanghai Sunred Biological Technology Co kits, China.
Diagnostic test: selected parameters of oxidative stress - carboxymethyle(lysine) (CML) | 3 years
  Serum concentration of carboxymethyle(lysine) (CML) [µg/mg protein] was determined with the enzyme immunoassay method (ELISA) for CML using Shanghai Sunred Biological Technology Co kits, China.
Diagnostic test: selected parameters of oxidative stress - advanced oxidation protein products (AOPP) | 3 years
  Serum concentration of advanced oxidation protein products (AOPP) [µmol/mg protein] was determined with the enzyme immunoassay method (ELISA) for AOPP using Shanghai Sunred Biological Technology Co kits, China.
Diagnostic test: metalloproteinases - metalloproteinase 9 (MMP-9) | 3 years
  metalloproteinase 9 (MMP-9) [ng/ml] concentration in the serum was determined by the ELISA method using the Quantikine Human MMP-9 (total) kit, by R&D Systems, Canada.
Diagnostic test: metalloproteinases - tissue inhibitor of metalloproteinase 1 (TIMP-1) | 3 years
  tissue inhibitor of metalloproteinase 1 (TIMP-1) [ng/ml] concentration in the serum - was determined by the ELISA method using the Quantikine Human TIMP-1 kit, manufactured by R&D Systems, Canada.
The MMP-9/TIMP-1 ratio assessment | 3 years
  the MMP-9/TIMP-1 ratio was calculated by the quotient of the MMP-9 [ng/ml] and the TIMP-1 [ng/ml] concentration.
Diagnostic test: selected inflammatory markers - high-sensivity C-reactive protein (hsCRP) | 3 years
  high-sensitivity C-reactive protein (hsCRP) [mg/l] concentration in the serum was measured using DADE Behring, USA, and the DADE nephelometer Behring Analyzer II.
Diagnostic test: selected inflammatory markers - neopterin | 3 years
  neopterin [nmol/l] serum concentration was determined by using the Neopterin ELISA kit, DRG International, Inc., USA.
Diagnostic Test: selected inflammatory markers - interleukin 18 (IL-18) | 3 years
  interleukin 18 (IL-18) [pg/ml] concentration in the serum was determined by Colorimetric Sandwich ELISA, Quantikine Human IL-18 R&D Inc., USA.
Diagnostic test: selected parameters of oxidative stress - myeloperoxidase (MPO) | 3 years
  myeloperoxidase (MPO) [ng/ml] in the serum - was determined by the ELISA method using the Quantikine Human MPO test by R&D Systems kit, Canada.
Diagnostic test: selected parameters of oxidative stress - methylglyoxal (MG) | 3 years
  methylglyoxal (MG) [µg/mg protein] concentration in the serum was assessed by competitive enzyme immunoassay (competitive ELISA) using MG kits from Cell Biolabs Inc, USA.
Diagnostic test: selected parameters of oxidative stress - carboxyethyle(lysine) (CEL) [µg/mg protein] | 3 years
  carboxyethyle(lysine) (CEL) [µg/mg protein] concentration in the serum was assessed by competitive enzyme immunoassay (competitive ELISA) using CEL kits from Cell Biolabs Inc, USA.
Diagnostic test: selected parameters of oxidative stress - carbamyl protein groups [µg/mg protein] | 3 years
  carbamyl protein groups [µg/mg protein] concentration in the serum were assessed by competitive enzyme immunoassay (competitive ELISA) using carbamyl protein groups kits from Cell Biolabs Inc, USA.
Diagnostic test: selected parameters of oxidative stress - soluble receptor for advanced glycation end products (sRAGE) | 3 years
  soluble receptor for advanced glycation end products (sRAGE) [µg/mg protein] concentration in the serum was tested with enzymatic immunoassay (Quantikine ELISA) using R&D Systems sRAGE kit, Canada.
Non-invasive cardiological examinations (1) with the use of Portapres device (Finapres Medical Systems (FMS), the Netherlands), the SphygmoCor tonometer (AtCor Medical), the Colin blood pressure monitor (BMP)-7000 (Japan) - blood pressures | 3 years
  Blood pressure was measured using the Colin BPM 7000 on both arms (participants were seated). Next, a piezoelectric tonometer Colin BPM was placed over the radial artery for the acquisition of the radial arterial pressure waveform in a supine position. This signal was sent to the SphygmoCor and after averaging various parameters have been assessed and recorded:
  * peripheral systolic blood pressure (sSBP) [mmHg];
  * peripheral diastolic blood pressure (pDBP)[mm Hg];
  * peripheral mean arterial pressure (pMAP) [mm Hg];
  * peripheral end-systolic pressure (pESP) [mm Hg];
  * central systolic blood pressure (cSBP) [mm Hg];
  * central diastolic blood pressure (cDBP) [mm Hg];
  * central mean arterial pressure (cMAP) [mm Hg];
  * entral augmented pressure (cAP) [mm Hg];
  * central mean pressure of diastole (cMPD) [mm Hg];
  * central mean pressure of systole (cMPS)[mm Hg];
  * central end-systolic pressure (cESP)[mm Hg]
Non-invasive cardiological examinations (2) with the use of Portapres device (Finapres Medical Systems (FMS), the Netherlands), the SphygmoCor tonometer (AtCor Medical), the Colin blood pressure monitor (BMP)-7000 (Japan) - heart rate (HR) | 3 years
  Blood pressure was measured using the Colin BPM 7000 on both arms (participants were seated). Next, a piezoelectric tonometer Colin BPM was placed over the radial artery for the acquisition of the radial arterial pressure waveform in a supine position. This signal was sent to the SphygmoCor and after averaging various parameters have been assessed and recorded:
  - heart rate (HR) in beats per minute [bpm]
Non-invasive cardiological examinations (3) with the use of Portapres device (Finapres Medical Systems (FMS), the Netherlands), the SphygmoCor tonometer (AtCor Medical), the Colin blood pressure monitor (BMP)-7000 (Japan) - ejection duration (ED) | 3 years
  Blood pressure was measured using the Colin BPM 7000 on both arms (participants were seated). Next, a piezoelectric tonometer Colin BPM was placed over the radial artery for the acquisition of the radial arterial pressure waveform in a supine position. This signal was sent to the SphygmoCor and after averaging various parameters have been assessed and recorded:
  - ejection duration (ED) in milliseconds [msec]
Device: carotid intima-media thickness (IMT) | 3 years
  Carotid intima-media thickness (IMT) [mm] was measured by The Accuson CV 70 system (Siemens) with a 10 megahertz (Mhz) transducer.
  Two longitudinal projections were assessed (anterolateral and posterolateral). The distal 1 cm of the common carotid artery just proximal to the bulb was measured by means of a computer analysis system (Medical Imaging Applications, LLC).
Device: vessel stiffness assessments - reflection index (RI) | 3 years
  The following parameter of vessel stiffness was assessed by Pulse Trace 2000 (Micro Medical Ltd., Rochester, Kent, United Kingdom):
  - reflection index (RI) in percentages [%].
Device: vessel stiffness assessments - vascular stiffness index (SI) | 3 years
  The following parameter of vessel stiffness was assessed by Pulse Trace 2000 (Micro Medical Ltd., Rochester, Kent, United Kingdom):
  -vascular stiffness index (SI) [m/s].
Device: vessel stiffness assessments - peripheral (pPP) and central pulse pressure (cPP) [mm Hg] | 3 years
  The following parameters of vessel stiffness were assessed by Pulse Trace 2000 (Micro Medical Ltd., Rochester, Kent, United Kingdom):
  * peripheral pulse pressure (pPP) [mm Hg];
  * central pulse pressure (cPP) [mm Hg]
Device: vessel stiffness assessments - peripheral pulse pressure/central pulse pressure (pPP/cPP) ratio | 3 years
  Peripheral pulse pressure/central pulse pressure (pPP/cPP) ratio was assessed by dividing peripheral pulse pressure (pPP) [mm Hg] by central pulse pressure (cPP) [mm Hg].
Cardiovascular (CV)-related death recording during 2-year follow-up | 2 years for each person qualified for the study
  During a 2-year follow-up from the enrollment to this study, CV-related fatal incidents history has been recorded for each subject separately. The primary endpoint was fatal acute myocardial infarction (AMI) or acute ischemic stroke or any unexpected or sudden death only if autopsy proved CV-related. If there was doubt about the cause of death or there was no contact with the patient during the two years from study enrollment, that patient was excluded and not considered further.
Diagnostic test: N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 3 years
  N-terminal pro-B-type natriuretic peptide (NT-proBNP) [fmol/ml] concentration in the serum was analyzed by enzyme immunoassay using the Nt-proBNP kit from Biomedica, Slovakia.

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Formanowicz, MD, PhD, Principal Investigator — Poznan University of Mediccal Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

REFERENCES:
- [Derived] Twardawa M, Formanowicz P, Formanowicz D. Chronic Kidney Disease as a Cardiovascular Disorder-Tonometry Data Analyses. Int J Environ Res Public Health. 2022 Sep 28;19(19):12339. doi: 10.3390/ijerph191912339. PMID 36231682
- [Derived] Kasprzak L, Twardawa M, Formanowicz P, Formanowicz D. The Mutual Contribution of 3-NT, IL-18, Albumin, and Phosphate Foreshadows Death of Hemodialyzed Patients in a 2-Year Follow-Up. Antioxidants (Basel). 2022 Feb 11;11(2):355. doi: 10.3390/antiox11020355. PMID 35204237